CLINICAL TRIAL: NCT04824378
Title: Study on Classification Method of Indocyanine Green Lymphography in Diagnosing Breast Cancer-related Lymphedema Based on Deep Learning
Brief Title: Study on Classification Method of Indocyanine Green Lymphography Based on Deep Learning
Acronym: BCRL；ICG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKUPH202102
Record Dates: First submitted 2021-03-27; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Breast Cancer Related Lymphedema; Deep Learning
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- label 1: Baseline data measurement of this group of patients: arm circumference（positive） and ICG (positive).
  Interventions: Other: No Intervention.
- label 2: Baseline data measurement of this group of patients: arm circumference（negative） and ICG (positive).
  Interventions: Other: No Intervention.
- label 3: Baseline data measurement of this group of patients: arm circumference（negative） and ICG (negative).
  Interventions: Other: No Intervention.

INTERVENTIONS:
Other: No Intervention. — No Intervention.Only learn ICG image features of different label groups

SUMMARY:
Breast cancer related lymphedema (BCRL) is the most common complication after breast cancer surgery, which brings a heavy psychological and spiritual burden to patients. For a long time, the diagnosis and treatment of lymphedema has been a difficult point in domestic and foreign research. To a large extent, it is because most of the patients who come to see a doctor have already developed obvious lymphedema, and the internal lymphatic vessels have undergone pathological remodeling[1] Therefore, it is particularly important to detect early lymphedema and intervene in time through the use of sensitive screening tools. Indocyanine green (ICG) lymphangiography is a relatively new method, which can display superficial lymph flow in real time and quickly, and will not be affected by radioactivity [7]. In 2007, indocyanine green lymphography was used for the first time to evaluate the function of superficial lymphatic vessels. In 2011, Japanese scholars found skin reflux signs based on ICG lymphography data of 20 patients with lymphedema after breast cancer surgery, and they were roughly divided into three types according to their severity: splash, star cluster, and diffuse (Figure 1) [8]. Later, in 2016, a prospective study involving 196 people affirmed the value of ICG lymphography in the early diagnosis of lymphedema, and made the images of ICG lymphography more specific stages 0-5 [9], but The staging is still based on the three types of skin reflux symptoms found in a small sample clinical study in 2011, which is not completely applicable in actual clinical applications. In addition, when abnormal skin reflux symptoms appear on ICG lymphangiography, the pathophysiological changes that occur in the body lack research and exploration. Therefore, this research hopes to refine the image features of ICG lymphography through machine learning (deep learning), and establish a PKUPH model for diagnosing early lymphedema by staging the image features.

ELIGIBILITY:
Inclusion Criteria:

* From October 2016 to present, about 200 patients who have been admitted to the Breast Surgery Clinic due to the main complaint of upper extremity edema, are willing to accept ICG lymphography, arm circumference measurement, drainage measurement, bioelectrical impedance measurement, main complaint scale, etc. .

Exclusion Criteria:

* Bilateral breast cancer; history of contrast agent allergy; arteriovenous thrombosis in the affected limb; regional lymph node recurrence; no informed consent; severe heart and brain diseases; primary lymphatic system disease (such as lymphatic leakage); unilateral only The limbs received ICG imaging.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients who have been admitted to the Breast Surgery Clinic due to the main complaint of upper extremity edema
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Establish a PKUPH model for the diagnosis of lymphedema by ICG based on deep learning | 2016-2022
  Establish a PKUPH model for the diagnosis of lymphedema by ICG based on deep learning

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, Dr, Principal Investigator — Breast Center, Peking University People's Hospital, Beijing, China
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
there is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Beek MA, te Slaa A, van der Laan L, Mulder PG, Rutten HJ, Voogd AC, Luiten EJ, Gobardhan PD. Reliability of the Inverse Water Volumetry Method to Measure the Volume of the Upper Limb. Lymphat Res Biol. 2015 Jun;13(2):126-30. doi: 10.1089/lrb.2015.0011. PMID 26091408
- [Background] Shi S, Lu Q, Fu MR, Ouyang Q, Liu C, Lv J, Wang Y. Psychometric properties of the Breast Cancer and Lymphedema Symptom Experience Index: The Chinese version. Eur J Oncol Nurs. 2016 Feb;20:10-6. doi: 10.1016/j.ejon.2015.05.002. Epub 2015 Jun 9. PMID 26071198
- [Background] Mihara M, Hara H, Araki J, Kikuchi K, Narushima M, Yamamoto T, Iida T, Yoshimatsu H, Murai N, Mitsui K, Okitsu T, Koshima I. Indocyanine green (ICG) lymphography is superior to lymphoscintigraphy for diagnostic imaging of early lymphedema of the upper limbs. PLoS One. 2012;7(6):e38182. doi: 10.1371/journal.pone.0038182. Epub 2012 Jun 4. PMID 22675520
- [Background] Yamamoto T, Yamamoto N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. Indocyanine green-enhanced lymphography for upper extremity lymphedema: a novel severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 Oct;128(4):941-947. doi: 10.1097/PRS.0b013e3182268cd9. PMID 21681123